CLINICAL TRIAL: NCT05972772
Title: A Pharmacokinetic-pharmacodynamic Study of Early Rickettsia Clearance in Murine Typhus or Scrub Typhus Patients Treated with Doxycycline or Azithromycin
Brief Title: Rickettsia Clearance Study
Acronym: RiCS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26-23
Record Dates: First submitted 2023-06-07; First posted 2023-08-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infectious Disease; Therapeutics
Keywords: Scrub Typhus; Typhus, Endemic Flea-Borne
MeSH Terms: conditions — Communicable Diseases; Scrub Typhus; Typhus, Endemic Flea-Borne | interventions — Doxycycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline (Active Comparator): Doxycycline (Vibramycin, 100-mg film-coated tablets; Pfizer)) 200-mg loading dose, followed by 100 mg every 12 hours for 3 days.
  Interventions: Drug: Doxycyclin
- Azithromycin (Active Comparator): Azithromycin (Zithromax, 250-mg capsules; Pfizer) with a 500-mg loading dose, followed by 250 mg every 24 hours for 2 days. This will be followed by three days of doxycycline at the dose in A.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Doxycyclin — 100-mg film-coated tablets; Pfizer
  Other Names: vibramycin
  Arms: Doxycycline
Drug: Azithromycin — 250-mg capsules; Pfizer
  Other Names: Zithromax
  Arms: Azithromycin

SUMMARY:
Murine typhus is a disease caused by Rickettisa typhi, an obligate intracellular bacterium transmitted by rodent fleas. The disease has a worldwide distribution; however the true burden is unknown, related to its non-specific presentation and lack of access to diagnosis in many regions. A systematic review of untreated murine typhus based on observational studies of a total of 239 patients has estimated the mortality associated with the disease at between 0.4% and 3.6%.

Scrub typhus is caused by Orientia tsutsugamushi and transmitted by the larval stage of chigger mites (Trombiculidae family). It has been estimated to affect at least one million people each year. A systematic review found varying reports of the mortality associated with untreated scrub typhus ranging from 0-70% (median 6%).

Polymerase chain reaction (PCR) based diagnosis of rickettsial infections is only available in one centre (Mahosot Hospital) in Vientiane. A number of hospitals use a variety of point-of-care antibody tests to diagnose rickettsial infections however many of these have not been validated and they are of uncertain sensitivity and specificity. In 2006 results of a two year prospective study of 427 patients presenting to Mahosot Hospital with a febrile illness and negative blood cultures showed that 115 (27%) patients had an acute rickettsial infection, confirmed by serological testing. Among these patients, 41 were diagnosed with murine typhus and 63 with scrub typhus. Antibacterial agents with activity against rickettsial pathogens include doxycycline, azithromycin, chloramphenicol and rifampicin. Azithromycin is often reserved for pregnant women or children below the age of 8 years due to lasting concerns after the tetracycline-associated staining of growing bones and teeth in the past. Evidence is accumulating that doxycycline is superior to azithromycin for the treatment of rickettsial disease. Clinical treatment failures have occurred following azithromycin treatment of murine typhus. The relationship between rickettsial bacteria load and both disease severity and response to treatment has not been characterised. Rickettsial concentrations in blood are generally low, of the order of 210 DNA copies/mL blood for R. typhi and 284 DNA copies/mL blood for O. tsutsugamushi. At present, there is no standard antibiotic susceptibility testing (AST) method for R. typhi and O. tsutsugamushi. The gold standard method for AST for Rickettsia pathogens is the plaque assay which determines minimal inhibitory concentration (MICs) from the smallest antimicrobial concentration inhibiting rickettsial plaque forming unit formation. This method is laborious and time consuming, taking approximately 14-16 days based on species to yield a result. Molecular detection methods are useful for diagnosing patients infected with rickettsial pathogens and has been applied for antibiotic susceptibility testing. Antibiotic susceptibility testing based on DNA synthesis inhibition detecting by quantitative PCR (qPCR) for O. tsutsugamushi clinical isolates has been reported. However, the relationship between antibiotic susceptibility profiles and treatment response has not been studied. There is a need to develop a reliable ex vivo method to characterize the treatment response and compare susceptibility of R. typhi and O. tsutsugamushi to different agents.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal 18 years
* Able to take oral medication
* Rapid test positive for murine typhus or scrub typhus
* Agrees to stay in hospital for at least 36 hours and to attend for scheduled follow up visits
* Written informed consent to participate in the study
* A negative urinary pregnancy test for all women of child-bearing age

Exclusion Criteria:

* Pregnancy or breast feeding
* Previous allergic reaction to doxycycline or azithromycin
* Received more than one dose of chloramphenicol, doxycycline, tetracycline, fluoroquinolones, rifampicin or azithromycin during this hospital admission or more than one dose of any of these drugs in the week before admission
* Contraindication to doxycycline: severe hepatic impairment, known SLE
* Contraindication to azithromycin: sever hepatic impairment
* Severe typhus defined as the presence of one or more of the following:

  1. Reduced level of consciousness
  2. Clinical jaundice
  3. Shock (BP systolic <80 mmHg)
  4. Unable to take oral medication
  5. Radiological evidence of pneumonia
  6. Clinical evidence for meningitis/encephalitis or the need of LP
  7. Alternative diagnosis confirmed that explains the presenting symptoms
  8. Any other syndrome which in the opinion of the admitting doctor constitutes severe typhus (reason must be stated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clearance of R. typhi or O. tsutsugamushi from peripheral blood of patients using serial qPCR measurement | Within 72 hours after treatment
  Measure of clearance or R. typhi or O. tsutsugamushi DNA assessed by serial qPCR measurements on the blood from murine typhus patients treated with either doxycycline or azithromycin. Rickettsia clearance rate will be estimated from serial qPCR measurement in each patient. The clearance rate is the slope of the initial log linear decline in qPCR estimated bacteria densities

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on plasma concentrations measure up to 96 hours after the last dose. Azithromycin: Based on plasma concentrations measure up to 2 weeks after the first dose.
  AUC of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Area under the intracellular concentration in the buffy coat versus time curve (AUC) of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on intracellular concentrations in the buffy coat measure up to 96 hours after the last dose. Azithromycin: Based on intracellular concentrations in Buffy coat measure up to 2 weeks after the first dose.
  AUC of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Peak plasma concentration (Cmax) of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on plasma concentrations measure up to 96 hours after the last dose. Azithromycin: Based on plasma concentrations measure up to 2 weeks after the first dose.
  Cmax of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Peak of the intracellular concentration (Cmax) in the buffy coat of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on intracellular concentrations in the buffy coat measure up to 96 hours after the last dose. Azithromycin: Based on intracellular concentrations in the buffy coat measure up to 2 weeks after the first dose.
  Cmax of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Time to peak plasma concentration (Tmax) of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on plasma concentrations measure up to 96 hours after the last dose. Azithromycin: Based on plasma concentrations measure up to 2 weeks after the first dose.
  Tmax of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Time to peak of the intracellular concentration (Tmax) in the buffy coat of doxycycline or azithromycin for the treatment of murine typhus or scrub typhus | Doxycycline: Based on intracellular concentrations in the buffy coat measure up to 96 hours after the last dose. Azithromycin: Based on intracellular concentrations in the buffy coat measure up to 2 weeks after the first dose.
  Tmax of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Time at doxycycline or azithromycin has lost half its maximum concentration (T1/2) for the treatment of murine typhus or scrub typhus | Doxycycline: Based on plasma concentrations measure up to 96 hours after the last dose. Azithromycin: Based on plasma concentrations measure up to 2 weeks after the first dose.
  T1/2 of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Time at doxycycline or azithromycin has lost half its maximum intracellular concentration (T1/2) for the treatment of murine typhus or scrub typhus | Doxycycline: Based on intracellular concentrations in the buffy coat measure up to 96 hours after the last dose. Azithromycin: Based on intracellular concentrations in the buffy coat measure up to 2 weeks after the first dose.
  T1/2 of doxycycline or azithromycin versus time from zero to infinity in the treatment of murine typhus and scrub typhus will be estimated using a modelling approach
Fever clearance time in patients with scrub typhus or murine typhus treated with doxycycline or azithromycin | First 7 days after treatment
  Fever clearance time is defined as the time in hours from onset of antibiotic treatment, to the first Axillary temperature recording less than or equal 37.5°C, which then remains less than or equal 37.5°C for 24 hours
Frequency of serious adverse events (SAEs) after treatment | Day 0 to day 28
  SAEs will be defined using the Common Toxicity Criteria (v5.0) of the US National Cancer Institute
Evaluation the accuracy of the new brand RDT, Rickettsia IgG/IgM Combo (Lumiquick) compared to Scrub typhus Detect IgM Rapid System (Dipstick) (InBios) | Day 0
  Sensitivity and specificity of Rickettsia IgG/IgM Combo (Lumiquick) compared to Scrub typhus Detect IgM Rapid System (Dipstick) (InBios) will be compared
Evaluation the accuracy of Rickettsia IgG/IgM Combo (Lumiquick) compared to a combined gold standard of PCR assays and serology (paired samples) | Day 0 and Day 28
  Sensitivity and specificity of RDT (Lumiquick) result will be compared to a combined gold standard of PCR assays and serology (paired serum)

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Phuklia, PhD, Principal Investigator — Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit
Locations (2):
- Laos (2):
  - Lao-Oxford-Mahosot Hospital-Wellcome Trust Research Unit (LOMWRU), Vientiane, Vientaine
  - Vientiane Provincial Hospital, Vientiane Province, Vientiane Province

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with data repositories or other researchers to use in the future.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: approximately 2 years after the end of the study